CLINICAL TRIAL: NCT07078149
Title: Knee Arthroplasty Surgery: Short-Term Effect of the ROSA Surgical Robot
Brief Title: Early Clinical Benefits of Robot-Assisted vs Manual Total Knee Arthroplasty (RATKA-EARLY)
Acronym: RATKA-EARLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Santa Cristina (Other)
Responsible Party: Principal Investigator, Inmaculada Neira, Orthopaedic surgeon, Hospital Universitario Santa Cristina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SantaCristinaH
Record Dates: First submitted 2025-06-19; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis (Knee OA); Total Knee Arthroplasty
Keywords: Robot-assisted total knee arthroplasty; ROSA Knee System; Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual TKA (mTKA) (Active Comparator): mTKA was performed using the conventional manual surgical technique, without robotic or navigation assistance. All bone cuts and implant positioning were carried out manually by the surgeon, based on preoperative planning and intraoperative anatomical landmarks. This approach represents the standard total knee arthroplasty technique widely used in routine clinical practice.
  Interventions: Procedure: Conventional manual TKA (mTKA)
- Robot-assisted TKA (RATKA) (Experimental): RATKA was performed using the ROSA® Knee System, a robotic-assisted surgical platform approved for total knee arthroplasty. The procedure was carried out by the surgeon with continuous manual control, while the robotic system provided intraoperative assistance to enhance the precision and reproducibility of bone resections and implant positioning.
  Interventions: Device: Robotic-assisted TKA (RATKA).

INTERVENTIONS:
Device: Robotic-assisted TKA (RATKA). — RATKA was performed using the ROSA® Knee System.
  Other Names: ROSA® Knee System
  Arms: Robot-assisted TKA (RATKA)
Procedure: Conventional manual TKA (mTKA) — mTKA was performed without robot assistance.
  Arms: Manual TKA (mTKA)

SUMMARY:
This study, called the RATKA-EARLY trial, was designed to compare two surgical techniques used in total knee replacement (also known as total knee arthroplasty or TKA). The aim was to determine whether the use of a robotic surgical system (ROSA® Knee System) offers short-term clinical advantages over the traditional manual technique.

A total of 68 adult patients with advanced knee osteoarthritis scheduled for TKA were enrolled. Participants were randomly assigned to one of two groups: 34 patients underwent robot-assisted TKA (RATKA), and 34 underwent conventional manual TKA (mTKA). All surgeries were performed by the same experienced surgical team, using the same type of implant.

Researchers assessed intraoperative and perioperative variables (such as surgical duration and blood loss), and evaluated early clinical outcomes at 3 months postoperatively by comparing pain levels, implant alignment, knee function, mobility, and overall patient satisfaction with baseline values.

The study was conducted at Hospital Universitario Santa Cristina in Madrid, Spain. It was approved by the local ethics committee and carried out in accordance with the Declaration of Helsinki and international research guidelines.

By comparing these two surgical approaches, the study aims to help patients and healthcare professionals make informed decisions regarding total knee replacement options.

DETAILED DESCRIPTION:
This was a prospective, randomized, controlled clinical trial including patients with knee osteoarthritis requiring total knee arthroplasty (TKA). Patients were randomized in a 1:1 ratio using a single-blind, parallel-group design based on a dice roll: even numbers assigned patients to the robot-assisted TKA (RATKA) group, and odd numbers assigned them to the conventional manual TKA (mTKA) group.

Inclusion criteria comprised symptomatic knee osteoarthritis with surgical indication for TKA and a correctable varus or valgus deformity of less than 18 degrees. Exclusion criteria included prior surgery on the index knee; prior arthroplasty in the same limb; neurological disorders affecting knee function; tumor involvement; ipsilateral hip pathology limiting range of motion (ROM); active periarticular infection; body mass index (BMI) > 35; dependency or institutionalization (e.g., nursing home residents); and severe anatomical deformity, instability, or malalignment requiring alternative surgical strategies.

Surgical procedures (RATKA using the ROSA® Knee System and mTKA) were performed as previously described in the literature. All surgeries were carried out by the same senior surgeon, who had previously completed the ROSA learning curve. A medial parapatellar approach and standard surgical exposure were used in all cases. The same posterior-stabilized implant design (Persona® PS; Zimmer Biomet, Warsaw, IN, USA) was implanted with patellar resurfacing and cement fixation (PALACOS® R+G, Heraeus). A tourniquet was placed but not inflated; no limb ischemia was induced. Tranexamic acid was administered intravenously unless contraindicated. Preoperative planning was based on full-length standing radiographs of the lower limbs (Tele-rx), and full-scale anteroposterior and lateral knee radiographs (AP/L-rx). Femoral and tibial osteotomies were calculated from mechanical axis measurements, and implant sizes were selected using AP/L-rx data. In the RATKA group, intraoperative registration was performed manually after arthrotomy, without the use of preoperative 3D imaging, in compliance with the Spanish Data Protection Act (Organic Law 3/2018). The ROSA® Knee System (software version 1.2; Zimmer Biomet) was used according to manufacturer guidelines.

The following data were collected. Baseline: demographic and clinical data (comorbidities, BMI, osteoarthritis severity using the Kellgren-Lawrence classification); hemoglobin and hematocrit values; radiographic studies (Tele-rx of the limb and AP/L knee views); and patient-reported outcome measures (PROMs) using the Visual Analog Scale (VAS) for pain, the Knee injury and Osteoarthritis Outcome Score (KOOS), and the 36-Item Short Form Health Survey (SF-36). Intraoperatively: operative time and intraoperative complications. Postoperative Day 3: hemoglobin and hematocrit values; radiographic studies (Tele-rx and AP/L views); functional recovery measured by range of motion (flexion and extension in degrees) using a goniometer; and mechanical limb alignment assessed on digital Tele-rx. Three months postoperatively: PROMs (VAS, KOOS, and SF-36); range of motion; radiographic studies (Tele-rx and AP/L views); and mechanical limb alignment measured again on digital Tele-rx.

Descriptive statistics were reported as frequencies for categorical variables and as means with standard deviations (SD) for continuous variables. Between-group comparisons were conducted using Student's t-tests or Mann-Whitney U tests for continuous variables, and chi-square or Fisher's exact tests for categorical variables. Pre- and postoperative clinical and radiographic outcomes were compared using paired t-tests or Wilcoxon signed-rank tests within groups, and unpaired t-tests or Mann-Whitney U tests between groups. Univariable and multivariable linear regression models were used to analyze VAS, KOOS, and SF-36 outcomes at 3 months. Multivariable models were adjusted for sex, age, BMI, and discharge values. All statistical analyses were performed using STATA 15 (StataCorp, College Station, TX, USA), with p-values < 0.05 considered statistically significant.

The study was approved by the Institutional Review Board of Hospital Universitario de La Princesa (Registry No. 4748; approval date: March 24, 2022). All procedures complied with the Declaration of Helsinki (2013 revision) and applicable Spanish regulations. Written informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee osteoarthritis with surgical indication for total knee arthroplasty (TKA)
* Correctable varus or valgus deformity of less than 18 degrees

Exclusion Criteria:

* Prior surgery on the index knee
* Prior arthroplasty in the same limb
* Neurological disorders affecting knee function
* Tumor involvement of the knee
* Ipsilateral hip pathology limiting range of motion (ROM)
* Active periarticular infection
* Body mass index (BMI) > 35
* Dependency or institutionalization (e.g., nursing home residents)
* Severe anatomical deformity, instability, or malalignment requiring alternative surgical strategies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Range of movement (ROM) | Baseline (before TKA) and three months after TKA.
  ROM (knee flexion and extension measured in degrees) was determined using a goniometer.
Pain intensity | From baseline (before TKA) to three months after TKA.
  Patient-reported outcome measure (PROM) of perceived pain intensity using the Visual Analog Scale (VAS; range: 0 to 10, where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate worse outcomes).
Knee injury and Osteoarthritis Outcome Score (KOOS) | From baseline (before TKA) to three months after TKA.
  Patient-reported outcome measure (PROM) using the full Knee injury and Osteoarthritis Outcome Score (KOOS), which includes five subscales: Pain, Symptoms, Activities of Daily Living (ADL), Sport and Recreation Function, and Knee-related Quality of Life (QOL). Each subscale score ranges from 0 to 100, where 0 indicates extreme problems and 100 indicates no problems. Higher scores represent better outcomes.
36-Item Short Form Health Survey (SF-36) | From baseline (before TKA) and three months after TKA.
  Patient-reported outcome measure (PROM) using the 36-Item Short Form Health Survey (SF-36), which assesses health-related quality of life across eight domains: Physical Functioning, Role Limitations due to Physical Health, Bodily Pain, General Health, Vitality (Energy/Fatigue), Social Functioning, Role Limitations due to Emotional Problems, and Mental Health. Scores for each domain range from 0 to 100, where 0 indicates the worst health status and 100 indicates the best possible health status. Higher scores represent better outcomes.
Blood loss | From baseline (before TKA) to hospital discharge (typically Day 3 post-TKA).
  Drop in hemoglobin and hematocrit values following TKA.
Operation time | During surgery.
  Duration of TKA
Mechanical alignment of the operated lower limb | Baseline (before TKA) and three months after TKA.
  Alignment was measured in degrees on digital Tele-rx.

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Neira, M.D., Principal Investigator — Hospital Universitario Santa Cristina
Locations (1):
- Hospital Universitario Santa Cristina, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning three months after publication and ending three years after the publication of results.
Access Criteria: De-identified individual participant data (IPD) will be shared with qualified researchers upon reasonable request after publication of the study results. Data will only be shared for purposes of academic, non-commercial research. Requests must include a clear description of the planned analyses. The proposed statistical methods may be subject to review by the original study team to ensure scientific integrity and appropriate use of the data.
  Researchers interested in accessing the data must submit a written proposal outlining the study objectives, planned analyses, and intended use. A data sharing agreement (DSA) must be signed to ensure data confidentiality and compliance with applicable regulations. Requests and documents can be submitted by email to the corresponding author after publication. Contact information will be provided in the published manuscript.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT07078149/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT07078149/ICF_001.pdf